CLINICAL TRIAL: NCT05845190
Title: Effect of Aerobic Training Versus Resistance Training on Plasma Homocystiene in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Egyptian Chinese University (Other)
Responsible Party: Principal Investigator, hanan hassan, Assistant lecturer, Egyptian Chinese University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P.T.REC/012/003654
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: simple randomization using a randomization table created by a computer software program
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercises group (group A ) (Experimental): 20 male patients with diabetes mellites Attended the program of walking on treadmill for 12 weeks according to the following parameters.
  Exercise prescription:
  Intensity: started by 60-75% of target heart rate according to each patient response.
  Duration: Each session consisted of five minutes warming up firstly then 25-30 minutes time of session ended by five minutes cool down exercises Frequency: Three times / week (day after day) for 12 weeks
  Interventions: Other: aerobic exercises
- resistance exercises group (group B) (Experimental): 20 male patients with diabetes mellites will participate in resistance training exercises 30-45 mins. The subject will warm up and cool down for at least five to seven minutes each, (before and after exercise) with initial load of 60% of 1 repetition maximum.
  This program consists of 3 sets of 8 to 12 repetitions, then increasing load when subject was able to complete 12 repetitions. A rest period of 1.5 min was established between each set.
  Mode: 4 upper body exercises (bench press, seated row, shoulder press, and pull down), 3 leg exercises (leg press, extension, and flexion), abdominal crunches and back extensions. with the individualized workloads at 60% of 1RM.
  Duration: 30 min-45 min (total session). Frequency: Three times / week (day after day). Intensity: increased load was established when subject was able to complete 12 repetitions.
  Interventions: Other: resistance exercises

INTERVENTIONS:
Other: aerobic exercises — aerobic exercises in form of walking on treadmill
  Other Names: group A
  Arms: aerobic exercises group (group A )
Other: resistance exercises — 60% of One-repetition maximum 3 sets ( 8 to 12 ) repetitions
  Other Names: group B
  Arms: resistance exercises group (group B)

SUMMARY:
The goal of this [clinical trial] is to [ compare ] in [ diabetic male patients ]. The main question to answer is :

Will be any difference between aerobic exercises and resistance exercises in improving levels of homocysteine, cholesterol and insulin in diabetic patients?

Participants will take their medications and group of them do aerobic exercises and another group do resistance training

DETAILED DESCRIPTION:
40 male diabetic patients diagnosed by type 2 diabetes mellites to evaluate therapeutics outcomes of aerobic exercises versus resistance exercises as a treatment tool on homocysteine, insulin and cholesterol levels in diabetic patients.

The patients will be randomly assigned to two equal (in number) groups:

Group (A) Twenty male patients will receive moderate intensity aerobic exercises in a form of supervised treadmill walking for 30-45 mins performed 3 times/ week for 12 weeks.

Group (B) Twenty male patients will receive resistance training program comprised 30-45 min performed 3 times /week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1- Their ages will range from 40 -55 years 2- Their body mass indexes will range between (25 to 35 Kg / m²). 3-All patients are diagnosed with type 2 diabetes mellites.
* Diagnostic criteria for type 2 diabetes were: 1) a fasting plasma glucose concentration of 7.0 mmol·L-1 or higher or 2) a plasma glucose concentration of 11.1 mmol·L-1 or higher two hours after an oral glucose challenge. (Punthakee et al.,2018).
* All subjects took oral hypoglycemic drugs but none of them were being treated with insulin when enrolled.

  4- All patients are medically and psychologically stable

Exclusion Criteria:

1. Patients with uncontrolled blood glucose level
2. Patients with unstable cardiovascular conditions (those with a known history of uncontrolled hypertension, ischemic attacks, stroke, congestive heart failure, currently on anticoagulation therapy) were excluded from this study.
3. Patients with severe pulmonary disease (with restrictive lung disease or with obstructive lung disease).
4. Patients with musculoskeletal disorders (Diagnosed with severe osteoporosis or severe osteoarthritis).
5. Patients with BMI > 35 will be excluded from the study.

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
homocystiene | 12 weeks of training
  Homocysteine was measured with an enzyme linked immunosorbent (ELISA) method. The upper limit of normal is 15 μmol/l

SECONDARY OUTCOMES:
insulin | 12 weeks of training
  normal value <25 mlu/L fasting
cholestrol | 12 weeks of trianing
  Desirable cholesterol levels are considered to be those below 200 mg/dL in adults

CONTACTS AND LOCATIONS:
Overall Officials: hanan hassan, Principal Investigator — Egyptian Chinese University
Locations (1):
- Egyptian Chineese University, Cairo, Gesr Elsuez, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all of the individual participant data collected during the trail, after de-identification
Time Frame: immediately following publication , no end data
Access Criteria: anyone who whishes to access the data, for any purpose